CLINICAL TRIAL: NCT07249372
Title: A Phase 2 Study of DRP-104, a Glutamine Antagonist, in Patients With NFE2L2/KEAP1-altered Non-Small Cell Lung Cancer
Brief Title: DRP-104 in Patients With NFE2L2/KEAP1-altered Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00948
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NFE2L2/KEAP1-Altered NSCLC (Experimental): Participants with NFE2L2/KEAP1-altered non-small cell lung cancer previously treated with chemotherapy and immunotherapy will receive subcutaneous DRP-104 (BIW) on a 21-day cycle with no rest period between cycles but with at least 3 days between injections.
  Interventions: Drug: DRP-104

INTERVENTIONS:
Drug: DRP-104 — DRP-104 will be administered subcutaneously (subQ) at a dose of 145mg twice a week (BIW) on a continuous schedule. Once the first dose is administered, the second weekly dose is to be administered 3 days after the first dose with a four-day rest period before the next week of therapy (example, Monday/Thursday or Tuesday/Friday).

SUMMARY:
This is a Phase 2 Study of DRP-104, a Glutamine Antagonist, in Patients with NFE2L2/KEAP1-altered Non-Small Cell Lung Cancer following standard of care treatment with chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* 18 years of age or older
* Diagnosis of advanced or recurrent, histologically or cytologically confirmed metastatic or unresectable non-small cell lung cancer harboring NFE2L2 or KEAP1 alterations
* Patients must have Response Evaluation Criteria in Solid Tumors (RECIST) measurable lesions
* At the time of enrollment, patients must have experienced progression of disease following treatment with standard of care chemotherapy and immune checkpoint inhibitors either sequentially or concurrently
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Patient should consent to allow the acquisition of existing Formalin-Fixed Paraffin-Embedded (FFPE) tumor tissue, as unstained slides, if available or to undergo a fresh tissue biopsy to obtain fresh tumor tissue for performance of correlative studies if deemed feasible. Tumor biopsies should only be performed if deemed safe and feasible by the investigator.
* Adequate baseline organ function:

  a) Absolute neutrophil count (ANC) ≥ 1.5x109/L (1500/uL);
* Without growth factor support for 7 days prior to screening labs for short acting growth factors and 14 days prior to screening labs for long-acting growth factors to meet eligibility
* b) Hemoglobin ≥ 9 g/dL
* Patients that require transfusion or growth factors need to demonstrate stable hemoglobin of ≥ 9 g/dL over at least a 7-day period after the last transfusion/growth factor injection prior to screening labs to meet eligibility)
* c) Platelets >75x109/L
* No transfusion 7 days prior to screening labs to meet eligibility
* d) Hepatic
* Total bilirubin ≤1.5 x upper limit of normal (ULN) or, in patients with Gilbert syndrome, total bilirubin >1.5 x ULN as long as direct bilirubin is normal
* PT/INR and PTT ≤1.5 x ULN, unless treated with anticoagulants
* AST(SGOT)/ALT(SGPT) ≤3 x ULN or ≤5 x ULN for patients with liver metastases/tumor infiltration
* e) Renal
* Adequate renal function as defined as Creatinine clearance ≥ 50 ml/min/1.73m2 measured or calculated by the Cockcroft-Gault equation or GFR ≥ 50 mL/min/1.73 m² by MDRD
* f) Cardiac
* Corrected QTc (Fridericia) < 470 ms
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use one highly effective method of contraception, including hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy or tubal ligation; and one effective method of contraception, including male condom, female condom, cervical cap, diaphragm or contraceptive sponge or abstain from heterosexual intercourse for the duration of study participation and for 5 half-lives of study drug plus 30 days (duration of ovulatory cycle) for a total of 5 weeks after completion of DRP-104. In addition, women must refrain from donating eggs during this time.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug plus 90 days (duration of sperm turnover) for a total of 14 weeks post completion of DRP-104. In addition, males must refrain from sperm donation during this time.
* Women must not be pregnant or breastfeeding or have intention of becoming pregnant during the study treatment or within for 5 half-lives of study drug plus 30 days (duration of ovulatory cycle) for a total of 5 weeks after completion of DRP-104.

Exclusion Criteria:

1. Target disease related criteria

   * Patients with progressive or symptomatic brain metastases will be excluded. Patients with brain metastases may be included in this trial as long as the brain metastases have completed definitive treatment at least 14 days prior treatment start and are radiologically stable (i.e., without evidence of progression on screening imaging assessment, [Note: repeat imaging should be performed during study screening]). Patients must be clinically stable and have discontinued anti-seizure medications and steroids, except for physiologic steroid dosing (≤10 mg/day of prednisone equivalents), for at least 14 days prior to Cycle 1 Day 1.
   * Any evidence of leptomeningeal disease
   * Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 8 weeks prior to Cycle 1 Day 1 and must have discontinued steroids, except for physiologic steroid dosing (≤10 mg/day of prednisone equivalents)
   * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently); Patients with indwelling catheters (e.g., PleurX) are allowed regardless of drainage frequency
2. Prior therapy

   * Patients who have not recovered to grade 1 or baseline from adverse events (CTCAE v 5.0) related to prior therapy excluding alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ grade 3. Lymphopenia ≤ grade 3 is allowed if not related to prior anticancer therapy. If related to prior anticancer therapy, lymphopenia must resolve to ≤ grade 1 or baseline.
   * Prior glutaminase inhibitor use
   * Prior systemic anticancer treatment (i.e., chemotherapy, biologic therapy [i.e., small molecular inhibitors], monoclonal antibodies, investigational agents]) within 21 days or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1. If a patient is receiving an anti-PD-1 or anti-PD-L1 antibody on a shorter frequency, i.e., every two weeks, then the patient is eligible if last dose is 14 days prior to Cycle 1 Day 1. Note: Patients must have recovered from all AEs due to previous therapies to CTCAE v 5.0 grade 1 or baseline, excluding, alopecia, peripheral neuropathy and ototoxicity, which must be at least grade 2 or baseline.
   * Prior palliative radiotherapy within 14 days prior to Cycle 1 Day 1 or within 42 days prior to Cycle 1 Day 1 from definitive local control radiation (any dose greater than 50 Gy, within 42 days of Cycle 1 Day1). Patients must have recovered from all radiation-related toxicities to CTCAE v 5.0 grade 1 or baseline, not require corticosteroids, and not have had radiation pneumonitis.
   * Prior therapy with long-acting myeloid growth factor or from a short acting myeloid growth factor within 14 days or 7 days prior to Cycle 1 Day 1, respectively
   * Any major surgery within 21 days prior to Cycle 1 Day 1 or who have not recovered from side effects of such procedure (CTCAE v 5.0 grade 1 or baseline)
   * Patients receiving potent inducers of CYP 3A4/5 (including St. John's Wort) that cannot be discontinued at least 14 days prior to Cycle 1 Day 1
3. Medical history and concurrent disease

   * Malignant disease, other than that being treated in this study. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Other exceptions include malignancies that were treated curatively and have not recurred within 3 years prior to Cycle 1 Day 1and any malignancy considered indolent and has never required therapy.
   * Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority
   * Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required during screening.
   * Impairment of gastrointestinal (GI) function or GI disease that may limit the ability to assess GI associated adverse events (e.g., ulcerative disease, uncontrolled nausea and diarrhea, vomiting, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
   * Uncontrolled concurrent illness including, but not limited to: ongoing or active infection; transfusion dependent thrombocytopenia or anemia that prevent meeting hematological inclusion criteria; psychiatric illness/social situations that would limit compliance with study requirements
   * Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following: Symptomatic congestive heart failure; Unstable angina pectoris or cardiac arrhythmia; Baseline corrected QTcF (Fridericia) ≥ 470 milliseconds; Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
   * A known or underlying medical condition that, in the opinion of the investigator or Sponsor, could make the administration of study drug/treatment hazardous to the patient, or could adversely affect the ability of the patient to comply with or tolerate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to Year 2
  ORR defined as the percentage of participants with a documented response [complete response (CR) or partial response (PR)] to the intervention.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to Year 2
  Measured as the time from first treatment with the intervention to date of first documented progression of disease - assessed among treated patients only.
Percentage of Patients with a Best Overall Response (BOR) of CR | Up to Year 2
Percentage of Patients with a Best Overall Response (BOR) of PR | Up to Year 2
Percentage of Patients with a Best Overall Response (BOR) of SD | Up to Year 2
Overall Survival (OS) | Up to Year 4
  OS measured as the time from first treatment with the intervention until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Punekar, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: salman.punekar@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to salman.punekar@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.